CLINICAL TRIAL: NCT05721729
Title: Phase 2 Crossover, Randomized, Placebo-Controlled, Single-Blind, Repeat Dose Study in Post-Bariatric Hypoglycemia Subjects to Determine the Effect of Mizagliflozin on Adverse Events and Postprandial Glucose Excursions
Brief Title: Effect of Mizagliflozin Repeat Dosing on Adverse Events and Postprandial Glucose Excursions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vogenx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VGX-001-012
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Postbariatric Hypoglycemia
MeSH Terms: interventions — mizagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Subjects will receive placebo and two doses of encapsulated mizagliflozin over three dosing periods. Once and twice daily dosing will be examined.
  Interventions: Drug: Mizagliflozin; Drug: Placebo
- Cohort 2 (Experimental): Subjects will receive placebo and two doses of encapsulated mizagliflozin over three dosing periods. Twice and three times daily dosing will be examined.
  Interventions: Drug: Mizagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Mizagliflozin — Encapsulated
Drug: Placebo — Encapsulated

SUMMARY:
This is a phase 2 crossover, randomized, placebo-controlled, single-blind, repeat dose study in PBH subjects to determine the effect of mizagliflozin on adverse events and postprandial glucose excursions.

DETAILED DESCRIPTION:
This is a phase 2 crossover, randomized, placebo-controlled, single-blind, repeat dose study in PBH subjects to determine the effect of mizagliflozin on adverse events and postprandial glucose excursions. This study will examine repeat doses of mizagliflozin and placebo while also evaluating dosing regimen. Up to 15 subjects are expected to complete the study. Subjects will be randomly assigned to a treatment arm within a cohort. Each subject should receive placebo and 2 active dose regimens in a crossover fashion.

ELIGIBILITY:
Inclusion Criteria:

* Roux-en-Y gastric bypass surgery performed > 6 months prior to enrollment
* Diagnosis of PBH

Exclusion Criteria:

* History of current medical conditions (other than PBH) which may result in hypoglycemia such as insulinoma, adrenal insufficiency, insulin autoimmune hypoglycemia, congenital hyperinsulinemia.
* Current use of insulin or insulin secretagogues
* History of current fasting hypoglycemia
* Pregnancy and/or lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 2 weeks after participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Through study completion, 43 days
  Number of participants with adverse events
Vital Signs | Through study completion, 43 days
  Number of participants with abnormal vital signs
Laboratory Tests | Through study completion, 43 days
  Number of participants with abnormal laboratory tests
Glucose nadir after dosing | 0-3 hours following liquid meal
  Time course of glucose concentrations during MMTT

SECONDARY OUTCOMES:
MMTT peak glucose concentration after dosing | 0-3 hours following liquid meal
  Time course of glucose concentrations during MMTT
MMTT peak insulin concentration after dosing | 0-3 hours following liquid meal
  Time course of insulin concentrations during MMTT
MMTT time to peak glucose concentration after dosing | 0-3 hours following liquid meal
  Time course of glucose concentrations during MMTT
MMTT time to peak insulin concentration after dosing | 0-3 hours following liquid meal
  Time course of insulin concentrations during MMTT
MMTT glucose concentration | 0-3 hours following liquid meal
  MMTT glucose area under the curve (AUC0-1, AUC0-2, and AUC0-3) after dosing
MMTT insulin concentration | 0-3 hours following liquid meal
  MMTT insulin area under the curve (AUC0-1, AUC0-2, and AUC0-3) after dosing

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford, Palo Alto, California
  - University of Colorado / Anschutz Medical Campus, Aurora, Colorado